CLINICAL TRIAL: NCT01078818
Title: A Phase IV, Unicenter, Randomized, Double-Blind, Parallel-Group, Comparaty Study of Intravenous and Oral Iron vs Placebo in Patient Under Extracorporeal Circulation in Cardiovascular Surgery
Brief Title: Oral and Intravenous Iron in Patients Postoperative Cardiovascular Surgery Under Extracorporeal Circulation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Canaria Rafael Clavijo para la Investigación Biomédica (Other)
Responsible Party: Pilar Garrido Martin MD, Fundación Canaria Rafael Clavijo para la Investigación Biomédica
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Tratamiento con hierro/2007
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2010-03-03 (Estimated); Status verified 2007-05

CONDITIONS: Anaemia
Keywords: Cardiac surgery; Extracorporeal circulation; Anaemia; Intravenous iron; Oral Iron
MeSH Terms: conditions — Anemia | interventions — Ferric Oxide, Saccharated; ferrous fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- IV trivalent saccharose hydroxide ferrous (Experimental)
  Interventions: Drug: IV trivalent saccharose hydroxide ferrous
- Oral ferrous fumarate (Active Comparator)
  Interventions: Drug: Oral ferrous fumarate
- Oral and intravenous Placebo (Placebo Comparator)
  Interventions: Drug: Oral and intravenous Placebo

INTERVENTIONS:
Drug: IV trivalent saccharose hydroxide ferrous — Preoperative Period 5-10 days 200 mg Iron iv (Venofer® )in 200cc physiologic solution /24-48h x 3 dosis +1 oral placebo /24h Postoperative Period 1-3weeks 200 mg Iron iv (Venofer® )in 200cc physiologic solution/24-48h x 3 dosis + 1 oral placebo /24h One month Follow-up
  1 month 1 oral placebo /24h
  Other Names: Venofer
  Arms: IV trivalent saccharose hydroxide ferrous
Drug: Oral ferrous fumarate — 200cc physiologic solution iv placebo /24-48h x 3 dosis + 1 oral iron tablet/24h (Ferogradumet®)
  Postoperative Period:
  200cc physiologic solution iv placebo /24-48h x 3 dosis + 1 oral iron tablet/24h (Ferogradumet®) One month Follow-up: 1 oral iron tablet/24h Ferogradumet
  Arms: Oral ferrous fumarate
Drug: Oral and intravenous Placebo — Preoperative Period:1oral placebo/24h Postoperative Period:200cc physiologic solution iv placebo /24-48h x 3 dosis + 1oral placebo/24h One month Follow-up:1 oral placebo/24h
  Arms: Oral and intravenous Placebo

SUMMARY:
Anaemia is a common postoperative problem of cardiovascular surgery after cardiopulmonary bypass (CPB). Because of this the need for hemoderived blood transfusions is high. The purpose of this study was to compare the clinical efficacy of intravenous and oral iron in anaemia and the impact of the iron on the transfusion rate in postoperative cardiovascular surgery under extracorporeal circulation.

DETAILED DESCRIPTION:
Prospective double dummy triple blind study of 159 patients undergoing CPB; randomised in 3 groups treated with iron intravenously (iv) (group I), with iron orally (group II) controlled with placebo (group III). Patients from group I were treated with iv Iron sucrose , three doses of 100 mg of iv iron every 24 hours during postoperative hospitalization and 1 pill/24 h of oral placebo during the first month after discharge. Group II was programmed to receive 1 iron pill orally every 24 hours pre and postoperatively and up to one month after discharge and a placebo while hospitalized. Group III was programmed to receive an oral and iv placebo pre and postoperatively.

Variables were collected preoperatively, at operation room and at Intensive Care Unit admission and discharge, at postoperative floor discharge and at one month after surgical discharge.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age
* Patients subject to elective cardiac surgery under extracorporeal circulation
* Patients without previous anaemia, susceptible of treatment
* Patients without need of blood transfusion preoperative
* Patients providing written informed consent
* Patients who are able to complete all study visits per protocol

Exclusion Criteria:

* Patients subject to elective cardiac surgery, but without extracorporeal circulation
* Patients who were treated with fibrinolytic therapy 48 hours before the surgery
* Patients with history of impaired renal function, (e.g., calculated creatinine clearance <50 mL/min/1.73 m2)
* Patients operated of active endocarditis
* Redo-surgery patients
* Women who are pregnant or lactating
* Patients with clinical of digestive bleeding
* Patients with vitamin B12 deficit
* Patients with ferropenic anaemia
* Patients with clinical history of asthma or allergy
* Patients with active infection
* Patients who are included in another clinical study
* Patients with hepatic disease
* Patients with history of allergy to iron
* Patients unlikely to adhere to protocol follow-up

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2007-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Haemoglobin and Hematocrit values | 2 years
  The objective was to compare the clinical efficacy of intravenous and oral iron in anaemia and the impact on the transfusion rate needing in Cardiovascular surgery under cardiopulmonary bypass

SECONDARY OUTCOMES:
need for hemoderived blood transfusions, postoperative stay and hospital costs | 2 years
  The objective was to compare the clinical efficacy of intravenous and oral iron in anaemia and the impact on the transfusion rate needing in Cardiovascular surgery under cardiopulmonary bypass

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Garrido, MD, Study Director — Hospital Universitario de Canarias
Locations (1):
- Hospital Universitario de Canarias, Santa Cruz de Tenerife, Santa Cruz de Tenerife, Spain

REFERENCES:
- [Background] Reuler JB. Hypothermia: pathophysiology, clinical settings, and management. Ann Intern Med. 1978 Oct;89(4):519-27. doi: 10.7326/0003-4819-89-4-519. PMID 358883
- [Background] Huyzen RJ, van Oeveren W, Wei F, Stellingwerf P, Boonstra PW, Gu YJ. In vitro effect of hemodilution on activated clotting time and high-dose thrombin time during cardiopulmonary bypass. Ann Thorac Surg. 1996 Aug;62(2):533-7. PMID 8694618
- [Background] Kirklin JW. Open-heart surgery at the Mayo Clinic. The 25th anniversary. Mayo Clin Proc. 1980 May;55(5):339-41. No abstract available. PMID 6990115
- [Background] Chenoweth DE, Cooper SW, Hugli TE, Stewart RW, Blackstone EH, Kirklin JW. Complement activation during cardiopulmonary bypass: evidence for generation of C3a and C5a anaphylatoxins. N Engl J Med. 1981 Feb 26;304(9):497-503. doi: 10.1056/NEJM198102263040901. PMID 7453783
- [Background] Butler J, Rocker GM, Westaby S. Inflammatory response to cardiopulmonary bypass. Ann Thorac Surg. 1993 Feb;55(2):552-9. doi: 10.1016/0003-4975(93)91048-r. PMID 8431082
- [Background] Fuhrer G, Gallimore MJ, Heller W, Hoffmeister HE. Aprotinin in cardiopulmonary bypass--effects on the Hageman factor (FXII)--Kallikrein system and blood loss. Blood Coagul Fibrinolysis. 1992 Feb;3(1):99-104. doi: 10.1097/00001721-199202000-00014. PMID 1377956
- [Background] Boyle EM Jr, Lille ST, Allaire E, Clowes AW, Verrier ED. Endothelial cell injury in cardiovascular surgery: atherosclerosis. Ann Thorac Surg. 1997 Mar;63(3):885-94. doi: 10.1016/s0003-4975(97)00057-x. PMID 9066432
- [Background] Correction of the anemia of end-stage renal disease with recombinant human erythropoietin. N Engl J Med. 1987 Jul 23;317(4):249-51. doi: 10.1056/NEJM198707233170416. No abstract available. PMID 3600716
- [Background] Bracey AW, Radovancevic R, Riggs SA, Houston S, Cozart H, Vaughn WK, Radovancevic B, McAllister HA Jr, Cooley DA. Lowering the hemoglobin threshold for transfusion in coronary artery bypass procedures: effect on patient outcome. Transfusion. 1999 Oct;39(10):1070-7. doi: 10.1046/j.1537-2995.1999.39101070.x. PMID 10532600
- [Background] Fishbane S, Kowalski EA. The comparative safety of intravenous iron dextran, iron saccharate, and sodium ferric gluconate. Semin Dial. 2000 Nov-Dec;13(6):381-4. doi: 10.1046/j.1525-139x.2000.00104.x. PMID 11130261
- [Background] Rohling RG, Zimmermann AP, Breymann C. Intravenous versus oral iron supplementation for preoperative stimulation of hemoglobin synthesis using recombinant human erythropoietin. J Hematother Stem Cell Res. 2000 Aug;9(4):497-500. doi: 10.1089/152581600419161. PMID 10982248
- [Background] Madi-Jebara SN, Sleilaty GS, Achouh PE, Yazigi AG, Haddad FA, Hayek GM, Antakly MC, Jebara VA. Postoperative intravenous iron used alone or in combination with low-dose erythropoietin is not effective for correction of anemia after cardiac surgery. J Cardiothorac Vasc Anesth. 2004 Feb;18(1):59-63. doi: 10.1053/j.jvca.2003.10.012. PMID 14973801
- [Background] Goodnough LT, Skikne B, Brugnara C. Erythropoietin, iron, and erythropoiesis. Blood. 2000 Aug 1;96(3):823-33. PMID 10910892
- [Background] Andrews NC. Disorders of iron metabolism. N Engl J Med. 1999 Dec 23;341(26):1986-95. doi: 10.1056/NEJM199912233412607. No abstract available. PMID 10607817
- [Derived] Garrido-Martin P, Nassar-Mansur MI, de la Llana-Ducros R, Virgos-Aller TM, Rodriguez Fortunez PM, Avalos-Pinto R, Jimenez-Sosa A, Martinez-Sanz R. The effect of intravenous and oral iron administration on perioperative anaemia and transfusion requirements in patients undergoing elective cardiac surgery: a randomized clinical trial. Interact Cardiovasc Thorac Surg. 2012 Dec;15(6):1013-8. doi: 10.1093/icvts/ivs344. Epub 2012 Aug 31. PMID 22940889